CLINICAL TRIAL: NCT06304428
Title: Prevention of Injury in Skilled Nursing Facilities Through Optimizing Medications
Acronym: PRISM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Hebrew SeniorLife (Other); Brown University (Other); The American Health Care Association (Unknown); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Pro00114580
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Accidental Falls/Prevention and Control; Osteoporosis
Keywords: Osteoporosis; Deprescribing; Falls; Skilled Nursing Facilities
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deprescribing Care Model (Active Comparator): In this pragmatic, cluster randomized crossover trial 42 Skilled Nursing Facilities (SNF) will each receive 6 months of each care model in random sequence. All patients with OP fracture admitted to the SNF within the intervention time period will receive the full designated care model, even if their stay in the SNF extends into the next intervention period.
  Interventions: Other: Deprescribing Care Model
- Bone Heath Service Model (Active Comparator): In this pragmatic, cluster randomized crossover trial 42 Skilled Nursing Facilities (SNF) will each receive 6 months of each care model in random sequence. All patients with OP fracture admitted to the SNF within the intervention time period will receive the full designated care model, even if their stay in the SNF extends into the next intervention period.
  Interventions: Other: Bone Health Service Model
- Injury Prevention Service Model (Active Comparator): In this pragmatic, cluster randomized crossover trial 42 Skilled Nursing Facilities (SNF) will each receive 6 months of each care model in random sequence. All patients with OP fracture admitted to the SNF within the intervention time period will receive the full designated care model, even if their stay in the SNF extends into the next intervention period.
  Interventions: Other: Injury Prevention Service Model

INTERVENTIONS:
Other: Deprescribing Care Model — The Deprescribing Care Model is designed to deprescribe fall related medications (FRIDs)
  Arms: Deprescribing Care Model
Other: Bone Health Service Model — The Bone Health Service Model is designed to provide osteoporosis evaluation and management
  Arms: Bone Heath Service Model
Other: Injury Prevention Service Model — The Injury Prevention Service Model provides both the Deprescribing Care Model and the Bone Health Service Model.
  Arms: Injury Prevention Service Model

SUMMARY:
The goal of this clinical trial is to compare three care models for optimizing medications and preventing falls with broken bones in patients receiving rehabilitation after a hospitalization for a broken bone.

The primary outcome is injurious falls, with secondary outcomes measuring how the process of care is changed and capturing patient-reported outcomes valued by stakeholders.

The main questions this study aims to answer are:

* Which of the three models is more effective in preventing falls with fractures?
* What are the differences in patient-centered outcomes amongst the three models? These include pain, depression, anxiety, sleep, medication side effect burden, and fear of falling.
* What are the differences in osteoporosis treatment and medication burden?

The three care models are: a Deprescribing Care Model designed to reduce or stop fall-related medications, a Bone Heath Service Model designed to provide osteoporosis evaluation and management, and an Injury Prevention Service Model offering both services.

42 SNFs will participate in this study. The three models will be incorporated into the routine care of patients at these facilities who are receiving rehabilitation after a hospitalization for a fracture. All care models will be delivered remotely to patients in the SNF and after they transition home by a post-fracture nurse consultant supported by an interprofessional team.

This study has three aims. See Detailed Description for more details. This ClinicalTrials.gov record represents the Comparative Effectiveness Aim of the protocol.

DETAILED DESCRIPTION:
After hospitalization for fracture, approximately 60% of older adults receive post-acute care in Skilled Nursing Facilities (SNFs), but fewer than 20% of these individuals receive medication optimization, which is evidence-based care known to prevent additional injurious falls, fractures, and mortality. Therefore, there is an opportunity to substantially improve care and patient outcomes in this setting. The purpose of this study is to determine the comparative efficacy of a Deprescribing Care Model designed to deprescribe fall related medications (FRIDs), a Bone Heath Service Model designed to provide osteoporosis evaluation and management, or an Injury Prevention Service Model offering both services. All care models will be delivered remotely to patients in the SNF and after they transition home by a post-fracture nurse consultant supported by an interprofessional team. The primary outcome is injurious falls, with secondary outcomes measuring how the process of care is changed and capturing patient-reported outcomes valued by stakeholders.

Our Specific aims are to:

1. Conduct a randomized cluster crossover trial in fracture patients comparing the effectiveness of the Deprescribing Care Model, Bone Health Service Model, or Injury Prevention Service Model in 42 SNFs, with each SNF receiving 6 months of each intervention in random sequence. We will test for clinically important differences in patient-centered outcomes (living with medicines survey, PHQ-8 depression scale, anxiety, sleep, and pain scales) at 90 days and implementation measures osteoporosis prescriptions, drug burden) at the time of discharge.
2. Compare the effectiveness of the Deprescribing Care Model, Bone Health Service Model, or Injury Prevention Service Model on subsequent injurious fall and fractures for patients treated within the 42 randomized SNFs with those in 168 matched concurrent control SNFs. We will use data from the National Institute on Aging-funded Long-Term Care Data Cooperative which includes Minimum Data Set (MDS), Electronic Health Record (EHR), and Medicare (CMS) claims. To address decisional dilemmas, we will examine differences in efficacy by baseline estimated life expectancy and cognitive status.
3. Identify SNF characteristics associated with measures of effective model implementation. We hypothesize that organizational factors captured by SNF staff responses to surveys capturing organizational readiness for change will explain additional variance in implementation measures beyond factors known to be associated with care quality (staff turnover rates, for profit-status, region, case mix, and proportion of patients from racial and ethnic minority groups).

Study Design: In the Comparative Effectiveness Aim (Aim 1), we will conduct a pragmatic, cluster randomized crossover trial in 42 SNFs comparing the effectiveness of a Bone Health Service Model, a Deprescribing Care Model, or an Injury Prevention Service Model, all delivered remotely by a post-fracture nurse consultant supported by an interprofessional team. Every SNF will receive 6 months of each care model in random sequence. Follow-up for delivery of the care models will begin on the date that the first eligible patient from the facility is included in the study. All patients with osteoporotic (OP) fracture admitted to the SNF within the intervention time period will receive the full designated care model, even if their stay in the SNF extends into the next intervention period. One primary post-fracture nurse consultant will be assigned to each facility for the life of the study. To prevent contamination between models, the nurse consultant will double check the care model assigned before every patient/proxy encounter. Medication utilization (measured using EHR data) will be assessed at discharge and 90 days after SNF admission date, and Patient Reported Outcomes (PROs) (measured via survey) will be assessed at 90 days after SNF admission date, regardless of whether they have discharged home or remain in the SNF. We will therefore be able to compare the effectiveness of the models on important PROs, osteoporosis treatment rates, and FRID medication burden. Patients will be followed for injurious falls and fractures using administrative data and self-report during post-fracture nurse consultant calls until the end of the study period (up to 3 years, mean 2 years) censoring at death.

In the Overall Effectiveness Aim, we will compare rates of injurious falls and fractures for patients treated with the Deprescribing Care Model, Bone Health Service Model, or Injury Prevention Service Model to patients treated in 168 matched concurrent control SNFs, identified through the Long Term Care Data Cooperative. No new data will be collected for this aim.

In the Implementation Evaluation Aim, we will identify facility characteristics associated with high levels of intervention implementation. This aim will require the collection of surveys from facility leadership.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or greater
* Admitted to an enrolled SNF after hospitalized fracture
* Completion of a medication optimization plan

Exclusion Criteria:

* Non-osteoporotic fracture (e.g. facial, digital, skull, at site of tumor or infection)
* Eligible for Hospice or palliative care
* Patient discharged or died prior to completion of a medication optimization plan

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3780 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Injurious falls | Up to 3 years
  Composite outcome of unique claims for emergency department, urgent care, or hospital visit for injurious fall or any fracture during follow-up (up to 3 years) (ICD 10 codes); to ensure complete ascertainment for participants with Medicare Advantage, researchers will also collect via self-report/proxy report at telephone calls 1, 3, 6, 12, 18 months, and 24 months following discharge from the SNF.

SECONDARY OUTCOMES:
Number of patients who initiate treatment for osteoporosis | 1 day of discharge from SNF and one year
  Osteoporosis treatment (process outcome)
Medication Possession Ratio during follow-up, as measured by EHR and Medicare claims | Up to 3 years
  Osteoporosis treatment adherence (process outcome)
Number of patients who had deprescribing ordered | 1 day of discharge from SNF and 90 days after SNF admission date
  Fall-risk increasing drug (FRID) use (process outcome)
Modified Drug Burden Index during follow-up, as measured by EHR and Medicare claims | Up to 3 years
  Fall-risk increasing drug (FRID) use (process outcome)
Patient medication side effect burden, measured via Living with Medicines Questionnaire (LMQ3). | 90 days after SNF admission date
  The LMQ3 is a validated self-report questionnaire. Medication side effect burden is measured via composite scores ranging from: No burden at all (41-73); Minimal burden (74-106); Moderate burden (107-139); High burden (140-172); and Extremely high burden (173-205), as well as a visual analog scale with scores ranging from: no burden at all (0.0- 2.0); minimal burden (2.1 -4.0); moderate (4.1-5.9); high burden (6.0-7.9); extremely high burden (8.0-10.0).
Patient falls self-efficacy (i.e. fear of falling), measured via Falls Efficacy Scale | 90 days after SNF admission date
  The Falls Efficacy Scale is a validated self-report questionnaire. Scores range from 10-100. A total score of greater than 70 indicates that the person has a fear of falling.
Patient pain, measured via Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form | 90 days after SNF admission date
  The Pain Interference Short Form is a validated self-report questionnaire. Each item on the measure is rated on a 5-point scale (1=not at all; 2=a little bit; 3=somewhat; 4=quite a bit; and 5=very much) with a range in score from 6 to 30 with higher scores indicating a greater degree of pain interference.
Patient depression, measured via Patient Health Questionnaire survey (PHQ-8) | 90 days after SNF admission date
  The PHQ-8 is a validated questionnaire for assessing the severity of depression symptoms.The score for each item is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of: not at all, several days, more than half the days, and nearly every day, respectively. Total score for the 8 items ranges from 0 to 24. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Patient anxiety, measured via PROMIS anxiety short form survey | 90 days after SNF admission date
  The PROMIS anxiety short form survey is a validated self-report questionnaire. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety.
Patient sleep, measured via PROMIS sleep disturbance short form | 90 days after SNF admission date
  The PROMIS sleep disturbance short form is a validated self-report questionnaire. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen S Colon-Emeric, MD, MHS, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Marcus Institute for Aging Research, Hebrew SeniorLife, Boston, Massachusetts
  - Duke University School of Medicine, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry SD, Toles M, Travison TG, McConnell ES, Zullo AR, Little MO, Gwyther L, McDermott C, Lee R, Cary M, Syme M, Kissam S, Hecker E, MacLean KG, Colon-Emeric C. PReventing Injury in Skilled nursing facilities through optimizing Medications (PRISM), a protocol for a cluster randomized trial to reduce injurious falls in post-acute care. Trials. 2025 Sep 26;26(1):367. doi: 10.1186/s13063-025-09122-z. PMID 41013714